CLINICAL TRIAL: NCT01573195
Title: Implementation of Antimicrobial Stewardship and Decision Support Into the EPIC Electronic Medical Record
Brief Title: Merck IISP Stewardship Grant for Antibiotic Best Practices
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0168 (MSN141105); Merk Dr Fox (Other Grant/Funding Number: Proposal #38732)
Record Dates: First submitted 2011-05-04; First posted 2012-04-06 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Antibiotic Resistant Infection
Keywords: deescalation; best practice alert; antimicrobial stewardship

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All prescribing MDs at UWHC: Observational for accept, reject, or accept with modification of Best Practice Alers

SUMMARY:
The purpose of this study is to pilot the use of best practices alerts to enhance an antimicrobial stewardship program using the electronic medical record, EPIC.

DETAILED DESCRIPTION:
The purpose of this study is to pilot the use of best practices to enhance an antimicrobial stewardship program using the electronic medical record, EPIC. Screening information technology tools via SETNET/Safety SUrveyor(Premier) and the electronic anti-infective order form would allow for sufficient medical record review to create best practices alerts for the purpose of appropriate de-escalation of anti-invectives.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with prescribing privileges at the UWHC

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1285 consecutive patients issued BPA for de-escalation of antibiotics in EPIC
Sampling Method: Non-Probability Sample
Enrollment: 1285 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of best practice alerts(BPA) that were completely accepted, partially accepted, or rejected within 72 hours of issuing the BPA | One Year
  after issuing the BPA for deescalation, the responding healthcare provider will respond in one of the manners above

SECONDARY OUTCOMES:
The number and type of antiinfectives that were administered before and after(11days) the best practice alert is issued. | One year
  The antiinfective use before and after the BPA will be analyzed in detail. The number of antibiotics, percentage decrease(or less likely increase) in antiinfectives in the 3 days before BPA , and 11 days after the BPA will be analyzed. A cost analysis will be performed. Patient outcomes will not be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Barry C Fox, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospitals and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Schulz L, Osterby K, Fox B. The use of best practice alerts with the development of an antimicrobial stewardship navigator to promote antibiotic de-escalation in the electronic medical record. Infect Control Hosp Epidemiol. 2013 Dec;34(12):1259-65. doi: 10.1086/673977. Epub 2013 Oct 28. PMID 24225610